CLINICAL TRIAL: NCT01014091
Title: Safety and Immunogenicity Study of GSK Biologicals' Pandemic Influenza Candidate Vaccine (GSK2340272A) in Children Aged 3 to 9 Years
Brief Title: Study to Evaluate the Safety and Immunogenicity of GSK Biological Pandemic Candidate Influenza Vaccine (H1N1) in Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 113810
Record Dates: First submitted 2009-11-12; First posted 2009-11-16 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-05

CONDITIONS: Influenza
Keywords: influenza infection; GSK Bio's influenza vaccine GSK2340272A
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- GSK2340272A F1 Y3-5 GROUP (Experimental): Healthy male or female children, between 3 and 5 years of age (Y3-5) at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 1 (F1) in the deltoid region of the arm, according to a 0-21 day schedule.
  Interventions: Biological: GSK pandemic vaccine GSK2340272A
- GSK2340272A F1 Y6-9 GROUP (Experimental): Healthy male or female children, between 6 and 9 years of age (Y6-9) at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 1 (F1) in the deltoid region of the arm, according to a 0-21 day schedule.
  Interventions: Biological: GSK pandemic vaccine GSK2340272A
- GSK2340272A F2 Y3-5 GROUP (Experimental): Healthy male or female children, between 3 and 5 years of age (Y3-5) at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 2 (F2) in the deltoid region of the arm, according to a 0-21 day schedule.
  Interventions: Biological: GSK pandemic vaccine GSK2340272A
- GSK2340272A F2 Y6-9 GROUP (Experimental): Healthy male or female children, between 6 and 9 years of age (Y6-9) at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 2 (F2) in the deltoid region of the arm, according to a 0-21 day schedule.
  Interventions: Biological: GSK pandemic vaccine GSK2340272A
- GSK2340272A F3 Y3-5 GROUP (Experimental): Healthy male or female children, between 3 and 5 years of age (Y3-5) at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 3 (F3) in the deltoid region of the arm, according to a 0-21 day schedule.
  Interventions: Biological: GSK pandemic vaccine GSK2340272A
- GSK2340272A F3 Y6-9 GROUP (Experimental): Healthy male or female children, between 6 and 9 years of age (Y6-9) at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 3 (F3) in the deltoid region of the arm, according to a 0-21 day schedule.
  Interventions: Biological: GSK pandemic vaccine GSK2340272A

INTERVENTIONS:
Biological: GSK pandemic vaccine GSK2340272A — 2 intramuscular injections

SUMMARY:
The objective of this study is to evaluate the safety and immunogenicity study of GSK Biologicals' pandemic influenza candidate vaccine (GSK2340272A) in children aged 3 to 9 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* Children, male or female, aged between 3 and 9 years at the time of first study vaccination.
* Written informed consent obtained from the parent(s) or LAR(s) of the subject.
* Healthy children, as established by medical history and clinical examination when entering the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Clinically or virologically confirmed influenza infection within six months preceding the study start.
* Planned administration of any vaccine 30 days prior and 30 days after any study vaccine administration.
* Have received any seasonal flu vaccine since last year.
* Previous administration of any H1N1 A/California-like vaccine
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to enrolment in this study or planned administration during the study period. For corticosteroids, this will mean prednisone >= 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment:

  * Fever is defined as temperature >= 37.5°C on oral, axillary or tympanic setting, or >= 38°C on rectal setting.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned during the study.
* Any condition which, in the opinion of the investigator, renders the subject unfit for participation in the study.
* Child in Care.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-12-01; Primary Completion 2011-01-14 (Actual); Study Completion 2011-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Czechia (3):
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113810 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From a total of 60 subjects enrolled in the study only 58 were vaccinated.
Period: Overall Study
Arm/Group | GSK2340272A F1 Y3-5 Group | GSK2340272A F1 Y6-9 Group | GSK2340272A F2 Y3-5 Group | GSK2340272A F2 Y6-9 Group | GSK2340272A F3 Y3-5 Group | GSK2340272A F3 Y6-9 Group
Started | 7 | 13 | 5 | 15 | 6 | 12
Completed | 7 | 13 | 5 | 15 | 6 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2340272A F1 Y3-5 Group | GSK2340272A F1 Y6-9 Group | GSK2340272A F2 Y3-5 Group | GSK2340272A F2 Y6-9 Group | GSK2340272A F3 Y3-5 Group | GSK2340272A F3 Y6-9 Group | Total
Number analyzed (Participants) | 7 | 13 | 5 | 15 | 6 | 12 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.1 (0.9) | 7.5 (1.2) | 3.8 (0.84) | 7.3 (0.9) | 3.8 (0.98) | 7.6 (0.9) | 6.36 (1.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 2 | 4 | 1 | 3 | 20
  Male | 4 | 6 | 3 | 11 | 5 | 9 | 38

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against Vaccine H1N1 Antigen
Description: Humoral immune response in terms of vaccine H1N1 haemagglutination inhibition (HI) antibodies against A/California/7/2009 (H1N1)v-like virus (Flu A/CAL/7/09) has been assessed. Antibody titers were presented as geometric mean titers (GMTs).
Time Frame: At Day 42
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects who received 2 doses of study vaccine and for whom assay results were available for antibodies against H1N1 antigen for any blood sample taken up to Month 7 after first vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- GSK2340272A F1 Group: Healthy male or female children, between 3 and 9 years of age at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 1 (F1) in the deltoid region of the arm, according to a 0-21 day schedule.
- GSK2340272A F2 Group: Healthy male or female children, between 3 and 9 years of age at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 2 (F2) in the deltoid region of the arm, according to a 0-21 day schedule.
- GSK2340272A F3 Group: Healthy male or female children, between 3 and 9 years of age at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 3 (F3) in the deltoid region of the arm, according to a 0-21 day schedule.
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Titers | 954.6 [730 to 1248.4] | 838.1 [647 to 1085.5] | 359.1 [219.8 to 586.9]

2. Primary Outcome: Number of Seropositive Subjects for HI Antibodies
Description: A seropositive subject was defined as a subject with a serum HI titer equal to or above (≥) 1:10. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 42
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who received 2 doses of study vaccine and for whom assay results were available for antibodies against H1N1 antigen for any blood sample taken up to Month 7 after first vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Participants | 13 | 9 | 12

3. Primary Outcome: Number of Seroconverted Subjects in Terms of HI Antibodies
Description: Seroconversion (SCR) was defined as: For initially seronegative subjects [pre-vaccination titer below (<) 1:10], a post-vaccination titer ≥ 1:40. For initially seropositive subjects (pre-vaccination titer ≥ 1:10), at least a 4-fold increase in post-vaccination titer. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Participants | 13 | 9 | 12

4. Primary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer ≥ 1:40, which is usually accepted as indicating protection. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Participants | 13 | 9 | 12

5. Primary Outcome: Geometric Mean Fold Increase (GMFR) for Serum HI Antibody Titer
Description: GMFR, also called seroconversion factor (SCF), was defined as the fold increase in serum HI geometric mean titers (GMTs) post-vaccination compared to pre-vaccination. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Fold change | 64 [25.9 to 158.2] | 71.9 [24.4 to 212.1] | 40.3 [27 to 60.3]

6. Secondary Outcome: Number of Seropositive Subjects for HI Antibodies
Description: as for outcome 2
Time Frame: At Day 0, Day 21 and Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Participants
  Flu A/CAL/7/09, Day 0 | 6 | 3 | 4
  Flu A/CAL/7/09, Day 21 | 13 | 9 | 12
  Flu A/CAL/7/09, Month 7 | 13 | 9 | 12

7. Secondary Outcome: HI Antibody Titers Against Vaccine H1N1 Antigen
Description: as for outcome 1
Time Frame: At Day 0, Day 21 and Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Titers
  Flu A/CAL/7/09, Day 0 | 14.9 [6.9 to 32] | 11.7 [4.2 to 32.1] | 8.9 [4.9 to 16.2]
  Flu A/CAL/7/09, Day 21 | 429.1 [268.9 to 684.6] | 285.3 [137.7 to 591.1] | 123.2 [40.5 to 374.9]
  Flu A/CAL/7/09, Month 7 | 155.9 [104.1 to 233.6] | 108.7 [61.2 to 192.9] | 84.8 [53.7 to 134.1]

8. Secondary Outcome: Number of Seroconverted Subjects in Terms of HI Antibodies
Description: Seroconversion (SCR) was defined as: For initially seronegative subjects (pre-vaccination titer below < 1:10), a post-vaccination titer ≥ 1:40. For initially seropositive subjects (pre-vaccination titer ≥ 1:10), at least a 4-fold increase in post-vaccination titer. The flu strain assessed was Flu A/CAL/7/09.
Time Frame: At Day 21 and Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Participants
  Flu A/CAL/7/09, Day 21 | 13 | 8 | 9
  Flu A/CAL/7/09, Month 7 | 12 | 7 | 10

9. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies
Description: as for outcome 4
Time Frame: At Day 0, Day 21 and Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Participants
  Flu A/CAL/7/09, Day 0 | 6 | 2 | 2
  Flu A/CAL/7/09, Day 21 | 13 | 9 | 9
  Flu A/CAL/7/09, Month 7 | 13 | 8 | 11

10. Secondary Outcome: Geometric Mean Fold Increase (GMFR) for Serum HI Antibody Titer
Description: as for outcome 5
Time Frame: At Day 21 and Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | GSK2340272A F1 Group | GSK2340272A F2 Group | GSK2340272A F3 Group
Number analyzed (Participants) | 13 | 9 | 12
Fold change
  Flu A/CAL/7/09, Day 21 | 28.8 [16.4 to 50.5] | 24.5 [10 to 59.7] | 13.8 [7.2 to 26.5]
  Flu A/CAL/7/09, Month 7 | 10.5 [6 to 18.3] | 9.3 [3.6 to 23.9] | 9.5 [5.9 to 15.3]

11. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = incidence of a particular symptom regardless of intensity grade or relationship to vaccinations. Grade 3 pain (children below 6 years of age) = cried when limb was moved/spontaneously painful. Grade 3 pain (children above 6 years of age) = significant pain at rest; pain that prevented normal everyday activities. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects with at least 1 vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Y3-5 Group | GSK2340272A F1 Y6-9 Group | GSK2340272A F2 Y3-5 Group | GSK2340272A F2 Y6-9 Group | GSK2340272A F3 Y3-5 Group | GSK2340272A F3 Y6-9 Group
Number analyzed (Participants) | 7 | 13 | 5 | 15 | 6 | 12
Participants
  Any Pain, Dose 1 | 6 | 13 | 3 | 12 | 1 | 6
  Grade 3 Pain, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness, Dose 1 | 5 | 6 | 1 | 5 | 2 | 4
  Grade 3 Redness, Dose 1 | 0 | 1 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1 | 4 | 6 | 1 | 6 | 1 | 2
  Grade 3 Swelling, Dose 1 | 0 | 2 | 0 | 0 | 0 | 0
  Any Pain, Dose 2 | 5 | 12 | 3 | 12 | 1 | 4
  Grade 3 Pain, Dose 2 | 0 | 1 | 0 | 0 | 0 | 0
  Any Redness, Dose 2 | 4 | 6 | 2 | 4 | 3 | 4
  Grade 3 Redness, Dose 2 | 0 | 1 | 0 | 0 | 1 | 0
  Any Swelling, Dose 2 | 5 | 9 | 1 | 5 | 2 | 3
  Grade 3 Swelling, Dose 2 | 0 | 2 | 0 | 1 | 1 | 0
  Any Pain, Across doses | 6 | 13 | 4 | 13 | 2 | 6
  Grade 3 Pain, Across doses | 0 | 1 | 0 | 0 | 0 | 0
  Any Redness, Across doses | 5 | 9 | 3 | 8 | 3 | 7
  Grade 3 Redness, Across doses | 0 | 1 | 0 | 0 | 1 | 0
  Any Swelling, Across doses | 6 | 10 | 2 | 8 | 3 | 3
  Grade 3 Swelling, Across doses | 0 | 3 | 0 | 1 | 1 | 0

12. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = incidence of a particular symptom regardless of intensity grade or relationship to vaccinations. Grade 3 drowsiness = drowsiness which prevented normal everyday activities. Grade 3 irritability = crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite = not eating at all. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as causally related to the vaccination
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340272A F1 Y3-5 Group: Healthy male or female children, between 3 and 5 years of age at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 1 (F1) in the deltoid region of the arm, according to a 0-21 day schedule.
- GSK2340272A F2 Y3-5 Group: Healthy male or female children, between 3 and 5 years of age at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 2 (F2) in the deltoid region of the arm, according to a 0-21 day schedule.
- GSK2340272A F3 Y3-5 Group: Healthy male or female children, between 3 and 5 years of age at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 3 (F3) in the deltoid region of the arm, according to a 0-21 day schedule.
Arm/Group | GSK2340272A F1 Y3-5 Group | GSK2340272A F2 Y3-5 Group | GSK2340272A F3 Y3-5 Group
Number analyzed (Participants) | 7 | 5 | 6
Participants
  Any Drowsiness, Dose 1 | 3 | 2 | 3
  Grade 3 Drowsiness, Dose 1 | 0 | 0 | 0
  Related Drowsiness, Dose 1 | 0 | 0 | 0
  Any Irritability, Dose 1 | 2 | 2 | 0
  Grade 3 Irritability, Dose 1 | 0 | 0 | 0
  Related Irritability, Dose 1 | 0 | 0 | 0
  Any Loss of appetite, Dose 1 | 2 | 0 | 0
  Grade 3 Loss of appetite, Dose 1 | 0 | 0 | 0
  Related Loss of appetite, Dose 1 | 0 | 0 | 0
  Any Temperature, Dose 1 | 2 | 0 | 1
  Grade 3 Temperature, Dose 1 | 2 | 0 | 0
  Related Temperature, Dose 1 | 1 | 0 | 0
  Any Drowsiness, Dose 2 | 1 | 0 | 2
  Grade 3 Drowsiness, Dose 2 | 0 | 0 | 0
  Related Drowsiness, Dose 2 | 0 | 0 | 0
  Any Irritability, Dose 2 | 1 | 1 | 0
  Grade 3 Irritability, Dose 2 | 0 | 0 | 0
  Related Irritability, Dose 2 | 1 | 0 | 0
  Any Loss of appetite, Dose 2 | 1 | 0 | 0
  Grade 3 Loss of appetite, Dose 2 | 0 | 0 | 0
  Related Loss of appetite, Dose 2 | 0 | 0 | 0
  Any Temperature, Dose 2 | 0 | 0 | 1
  Grade 3 Temperature, Dose 2 | 0 | 0 | 0
  Related Temperature, Dose 2 | 0 | 0 | 0
  Any Drowsiness, Across doses | 4 | 2 | 3
  Grade 3 Drowsiness, Across doses | 0 | 0 | 0
  Related Drowsiness, Across doses | 0 | 0 | 0
  Any Irritability, Across doses | 3 | 2 | 0
  Grade 3 Irritability, Across doses | 0 | 0 | 0
  Related Irritability, Across doses | 1 | 0 | 0
  Any Loss of appetite, Across doses | 3 | 0 | 0
  Grade 3 Loss of appetite, Across doses | 0 | 0 | 0
  Related Loss of appetite, Across doses | 0 | 0 | 0
  Any Temperature, Across doses | 2 | 0 | 2
  Grade 3 Temperature, Across doses | 2 | 0 | 0
  Related Temperature, Across doses | 1 | 0 | 0

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal, headache and temperature [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)]. Any = incidence of a particular symptom regardless of intensity grade or relationship to vaccinations. Grade 3 = symptom which prevented normal everyday activity. Related = symptom assessed by the investigator as causally related to the vaccination. Grade 3 fever = fever > 39.0 °C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Groups:
- GSK2340272A F1 Y6-9 Group: Healthy male or female children, between 6 and 9 years of age at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 1 (F1) in the deltoid region of the arm, according to a 0-21 day schedule.
- GSK2340272A F2 Y6-9 Group: Healthy male or female children, between 6 and 9 years of age at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 2 (F2) in the deltoid region of the arm, according to a 0-21 day schedule.
- GSK2340272A F3 Y6-9 Group: Healthy male or female children, between 6 and 9 years of age at the time of first study vaccination, who intramuscularly received 2 doses of GSK2340272A vaccine formulation 3 (F3) in the deltoid region of the arm, according to a 0-21 day schedule.
Arm/Group | GSK2340272A F1 Y6-9 Group | GSK2340272A F2 Y6-9 Group | GSK2340272A F3 Y6-9 Group
Number analyzed (Participants) | 13 | 15 | 12
Participants
  Any Fatigue, Dose 1 | 5 | 5 | 8
  Grade 3 Fatigue, Dose 1 | 0 | 0 | 0
  Related Fatigue, Dose 1 | 3 | 0 | 2
  Any Gastrointestinal, Dose 1 | 3 | 2 | 2
  Grade 3 Gastrointestinal, Dose 1 | 0 | 0 | 0
  Related Gastrointestinal, Dose 1 | 1 | 0 | 0
  Any Headache, Dose 1 | 7 | 5 | 5
  Grade 3 Headache, Dose 1 | 0 | 0 | 0
  Related Headache, Dose 1 | 1 | 0 | 1
  Any Temperature/(Axillary), Dose 1 | 1 | 1 | 1
  Grade 3 Temperature/(Axillary), Dose 1 | 0 | 0 | 0
  Related Temperature/(Axillary), Dose 1 | 1 | 0 | 1
  Any Fatigue, Dose 2 | 6 | 7 | 1
  Grade 3 Fatigue, Dose 2 | 0 | 2 | 0
  Related Fatigue, Dose 2 | 2 | 2 | 1
  Any Gastrointestinal, Dose 2 | 4 | 3 | 0
  Grade 3 Gastrointestinal, Dose 2 | 0 | 0 | 0
  Related Gastrointestinal, Dose 2 | 2 | 0 | 0
  Any Headache, Dose 2 | 6 | 9 | 0
  Grade 3 Headache, Dose 2 | 1 | 1 | 0
  Related Headache, Dose 2 | 3 | 2 | 0
  Any Temperature/(Axillary), Dose 2 | 4 | 1 | 0
  Grade 3 Temperature/(Axillary), Dose 2 | 0 | 0 | 0
  Related Temperature/(Axillary), Dose 2 | 3 | 1 | 0
  Any Fatigue, Across doses | 6 | 9 | 8
  Grade 3 Fatigue, Across doses | 0 | 2 | 0
  Related Fatigue, Across doses | 3 | 2 | 3
  Any Gastrointestinal, Across doses | 4 | 3 | 2
  Grade 3 Gastrointestinal, Across doses | 0 | 0 | 0
  Related Gastrointestinal, Across doses | 2 | 0 | 0
  Any Headache, Across doses | 10 | 9 | 5
  Grade 3 Headache, Across doses | 1 | 1 | 0
  Related Headache, Across doses | 3 | 2 | 1
  Any Temperature/(Axillary), Across doses | 4 | 2 | 1
  Grade 3 Temperature/(Axillary), Across doses | 0 | 0 | 0
  Related Temperature/(Axillary), Across doses | 3 | 1 | 1

14. Secondary Outcome: Number of Subjects With Any Medically-attended Events (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: During the entire study period (from Month 0 up to Month 12)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Y3-5 Group | GSK2340272A F1 Y6-9 Group | GSK2340272A F2 Y3-5 Group | GSK2340272A F2 Y6-9 Group | GSK2340272A F3 Y3-5 Group | GSK2340272A F3 Y6-9 Group
Number analyzed (Participants) | 7 | 13 | 5 | 15 | 6 | 12
Participants | 4 | 11 | 5 | 11 | 6 | 10

15. Secondary Outcome: Number of Subjects With Adverse Events of Specific Interest (AESIs)/Potential Immune-mediated Disease (pIMDs)
Description: Adverse events of specific interest (AESI) were defined as AEs including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration. Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: During the entire study period (from Month 0 up to Month 12)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Y3-5 Group | GSK2340272A F1 Y6-9 Group | GSK2340272A F2 Y3-5 Group | GSK2340272A F2 Y6-9 Group | GSK2340272A F3 Y3-5 Group | GSK2340272A F3 Y6-9 Group
Number analyzed (Participants) | 7 | 13 | 5 | 15 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within the 42-day (Days 0-41) post-vaccination period
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Y3-5 Group | GSK2340272A F1 Y6-9 Group | GSK2340272A F2 Y3-5 Group | GSK2340272A F2 Y6-9 Group | GSK2340272A F3 Y3-5 Group | GSK2340272A F3 Y6-9 Group
Number analyzed (Participants) | 7 | 13 | 5 | 15 | 6 | 12
Participants
  Any AE(s) | 1 | 2 | 0 | 2 | 2 | 2
  Grade 3 AE(s) | 0 | 1 | 0 | 0 | 0 | 0
  Related AE(s) | 0 | 1 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 to Month 12)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2340272A F1 Y3-5 Group | GSK2340272A F1 Y6-9 Group | GSK2340272A F2 Y3-5 Group | GSK2340272A F2 Y6-9 Group | GSK2340272A F3 Y3-5 Group | GSK2340272A F3 Y6-9 Group
Number analyzed (Participants) | 7 | 13 | 5 | 15 | 6 | 12
Participants | 0 | 1 | 1 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period. Unsolicited adverse events (AEs): during the 21-day (Days 0-20) post-vaccination period. Serious adverse events (SAEs): from Month 0 up to Month 12.
Arm/Group | GSK2340272A F1 Y3-5 Group | GSK2340272A F1 Y6-9 Group | GSK2340272A F2 Y3-5 Group | GSK2340272A F2 Y6-9 Group | GSK2340272A F3 Y3-5 Group | GSK2340272A F3 Y6-9 Group
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/13 | 1/5 | 1/15 | 0/6 | 1/12
Other Adverse Events (participants affected / at risk) | 7/7 | 13/13 | 4/5 | 15/15 | 6/6 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2340272A F1 Y3-5 Group (N=7) | GSK2340272A F1 Y6-9 Group (N=13) | GSK2340272A F2 Y3-5 Group (N=5) | GSK2340272A F2 Y6-9 Group (N=15) | GSK2340272A F3 Y3-5 Group (N=6) | GSK2340272A F3 Y6-9 Group (N=12)
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2340272A F1 Y3-5 Group (N=7) | GSK2340272A F1 Y6-9 Group (N=13) | GSK2340272A F2 Y3-5 Group (N=5) | GSK2340272A F2 Y6-9 Group (N=15) | GSK2340272A F3 Y3-5 Group (N=6) | GSK2340272A F3 Y6-9 Group (N=12)
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 6 | 13 | 4 | 13 | 2 | 6
Redness (General disorders) | 5 | 9 | 3 | 8 | 3 | 7
Swelling (General disorders) | 6 | 10 | 2 | 8 | 3 | 3
Drowsiness (General disorders) | 4 | 0 | 2 | 0 | 3 | 0
Irritability (General disorders) | 3 | 0 | 2 | 0 | 0 | 0
Loss of appetite (General disorders) | 3 | 0 | 0 | 0 | 0 | 0
Temperature/(Axillary) (General disorders) | 2 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 6 | 0 | 9 | 0 | 8
Gastrointestinal (General disorders) | 0 | 4 | 0 | 3 | 0 | 2
Headache (General disorders) | 0 | 10 | 0 | 9 | 0 | 5
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4 | 0 | 2 | 4 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 2 | 1 | 1 | 2
Tonsillitis (Infections and infestations) | 0 | 4 | 1 | 2 | 0 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.